CLINICAL TRIAL: NCT01400867
Title: A Multicenter, Randomized, Observer-Blinded, Active-Controlled Study to Evaluate the Safety, Tolerability, Efficacy, and Pharmacokinetics of Ceftaroline Versus Comparator in Pediatric Subjects With Acute Bacterial Skin and Skin Structure Infections
Brief Title: Safety and Efficacy Study of Ceftaroline Versus a Comparator in Pediatric Subjects With Complicated Skin Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P903-23
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Infections, Pediatrics
Keywords: Infections; Pediatrics; Teflaro; cephalosporin
MeSH Terms: conditions — Infections | interventions — Ceftaroline; Cephalexin; Clindamycin; Linezolid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ceftaroline fosamil (Experimental)
  Interventions: Drug: Ceftaroline fosamil; Drug: Cephalexin or Clindamycin or Linezolid
- Comparators (Active Comparator): Vancomycin +/- Aztreonam Cefazolin +/- Aztreonam
  Interventions: Drug: Vancomycin +/- Aztreonam or Cefazolin +/- Aztreonam; Drug: Cephalexin or Clindamycin or Linezolid

INTERVENTIONS:
Drug: Ceftaroline fosamil — Subjects ≥ 6 months old: 12 mg/kg IV for subjects weighing ≤ 33 kg and 400 mg for subjects weighing > 33 kg will be infused over 60 (± 10) minutes every 8 hours (q8h) (± 1 hour)
  Subjects < 6 months old: 8mg/kg infused over 60 (± 10) minutes every 8 hours (q8h) (± 1 hour)
  Other Names: Teflaro; PPI-0903; TAK-599; TAK599; PPI0903
  Arms: Ceftaroline fosamil
Drug: Vancomycin +/- Aztreonam or Cefazolin +/- Aztreonam — Vancomycin 15mg/kg IV over 60 minutes (or a maximum of 10mg/min whichever is longer) +/- Aztreonam 30 mg/kg IV every 8 hours over 60 minutes (for infections involving gram negative pathogen suspected or confirmed)
  Cefazolin 75mg/kg IV divided every 8 hours over 60 minutes (for sites that do not empirically cover for MRSA) +/- Aztreonam 30 mg/kg IV every 8 hours over 60 minutes (for infections involving gram negative pathogen suspected or confirmed
  Arms: Comparators
Drug: Cephalexin or Clindamycin or Linezolid — Possible oral switch on or after study day 4.
  Cephalexin: 25 mg/kg q6h PO or Clindamycin: 10 mg/kg q8h PO or Linezolid 600mg q12h (cohort 1) or 10 mg/kg q8h (cohorts 2,3 and 4) PO.

SUMMARY:
This is a study of safety, effectiveness, blood levels and tolerance of Ceftaroline fosamil in children with skin infections receiving antibiotic therapy in the hospital.

DETAILED DESCRIPTION:
To evaluate safety, effectiveness, pharmacokinetics and tolerance of Ceftaroline fosamil in children who are initially hospitalized with Acute Bacterial Skin and Skin Structure Infections (ABSSSI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 2 months to < 18 years old.
* Presence of ABSSSI warranting initial hospitalization.
* Presence of ABSSSI with measurable margins of erythema, that includes deeper and/or extensive soft tissue involvement, or requires significant therapeutic surgical intervention

Exclusion Criteria:

* Documented history of any hypersensitivity or allergic reaction to vancomycin, aztreonam, or any β-lactam antimicrobial
* Uncomplicated skin and soft tissue infections
* More than 24 hours of prior antimicrobial therapy ≤ 96 hours before randomization.
* Requirement for any concomitant systemic antimicrobial therapy
* History of seizures, excluding well-documented febrile seizure of childhood.
* Clinical signs or suspicion of meningitis

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2011-12; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of ceftaroline versus comparator in pediatric subjects ages 2 months to < 18 years with ABSSSI. | Between 26 and 50 days.
  Evaluate the safety and tolerability of IV administered ceftaroline fosamil in children with skin infections. Summaries of AEs, SAEs, deaths, laboratory evaluations (hematology studies, comprehensive and metabolic panel), pain scales, vital signs, and physical examinations will be provided for each treatment group.

SECONDARY OUTCOMES:
Evaluate the efficacy of ceftaroline versus comparator in pediatric subjects ages 2 months to < 18 years with ABSSSI. | Between 1 and 5 days
  The number and percentage of subjects in each treatment group classified as clinical cure in the Modified Intent to Treat (MITT) and Clinical Evaluable (CE) populations at Day 3, EOIV, EOT and TOC.
Evaluate the pharmacokinetics of ceftaroline versus comparator in pediatric subjects ages 2 months to < 18 years with ABSSSI. | Between 1 and 5 days
  Analyze concentrations of ceftaroline fosamil, ceftaroline, and M-1 in plasma, and if available, in cerebrospinal fluid (CSF; if collected as part of routine medical care)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (28):
  - Investigational Site - Phoenix, Phoenix, Arizona
  - Investigational Site - Orange, Orange, California
  - Investigational Site - San Diego, San Diego, California
  - Investigational Site - Jacksonville, Jacksonville, Florida
  - Investigational Site - Atlanta, Atlanta, Georgia
  - Investigational Site - Chicago 1, Chicago, Illinois
  - Investigational Site - Chicago 2, Chicago, Illinois
  - Investigational Site - Springfield, Springfield, Illinois
  - Investigational Site - Shreveport, Shreveport, Louisiana
  - Investigational Site - Baltimore, Baltimore, Maryland
  - Investigational Site - Detroit, Detroit, Michigan
  - Investigational Site - Brooklyn, Brooklyn, New York
  - Investigational Site - New Hyde Park, New Hyde Park, New York
  - Investigational Site - Rochester, Rochester, New York
  - Investigational Site - Bronx, The Bronx, New York
  - Investigational Site - Akron, Akron, Ohio
  - Investigational Site - Cleveland 1, Cleveland, Ohio
  - Investigational Site - Cleveland 2, Cleveland, Ohio
  - Investigational Site - Toledo, Toledo, Ohio
  - Investigational Site - Pittsburgh, Pittsburgh, Pennsylvania
  - Investigational Site - Charleston, Charleston, South Carolina
  - Investigational Site - Memphis, Memphis, Tennessee
  - Investigational Site - Austin 1, Austin, Texas
  - Investigational Site - Fort Worth, Fort Worth, Texas
  - Investigational Site - Norfolk, Norfolk, Virginia
  - Investigational Site - Richmond, Richmond, Virginia
  - Investigational Site - Seattle, Seattle, Washington
  - Investigational Site - Morgantown, Morgantown, West Virginia
- Argentina (8):
  - Investigational Site - Buenos Aires 1, Buenos Aires
  - Investigational Site - Buenos Aires 2, Buenos Aires
  - Investigational Site - Buenos Aires 3, Buenos Aires
  - Investigational Site - Buenos Aires 4, Buenos Aires
  - Investigational Site - Buenos Aires 5, Buenos Aires
  - Investigational Site - Buenos Aires 6, Buenos Aires
  - Investigational Site - Santa Fe 1, Santa Fe
  - Investigational Site - Santa Fe 2, Santa Fe
- Chile (4):
  - Investigational Site - Puente Alto, Puente Alto, Santiago Metropolitan
  - Investigational Site - San Ramon, San Ramón, Santiago Metropolitan
  - Investigational Site - Vitacura, Vitacura, Santiago Metropolitan
  - Investigational Site - Vina Del Mar, Viña del Mar
- Georgia (2):
  - Investigational Site - Tbilisi 1, Tbilisi
  - Investigational Site - Tbilisi 2, Tbilisi
- Latvia (4):
  - Investigational Site - Daugavpils, Daugavpils
  - Investigational Site - Liepaja, Liepāja
  - Investigational Site - Rezekne, Rēzekne
  - Investigational Site - Riga, Riga
- Lithuania (2):
  - Investigational Site - Kaunas, Kaunas
  - Investigational Site - Vilnius, Vilnius
- Poland (6):
  - Investigational Site - Bydgoszcz 1, Bydgoszcz
  - Investigational Site - Bydgoszcz 2, Bydgoszcz
  - Investigational Site - Lodz, Lodz
  - Investigational Site - Lublin, Lublin
  - Investigational Site - Rzeszow, Rzeszów
  - Investigational Site - Warszawa, Warsaw
- Romania (5):
  - Investigational Site - Bucharest 1, Bucharest
  - Investigational Site - Bucharest 2, Bucharest
  - Investigational Site - Constanta, Constanța
  - Investigational Site - Tirgu Mures, Târgu Mureş
  - Investigational Site - Timisoara, Timișoara
- South Africa (4):
  - Investigational Site - Cape Town 1, Cape Town
  - Investigational Site - Cape Town 2, Cape Town
  - Investigational Site - Cape Town 3, Cape Town
  - Investigational Site - Johannesburg, Johannesburg
- Spain (8):
  - Investigational Site - Badalona, Badalona
  - Investigational Site - Esplugues de Llobregat, Esplugues de Llobregat
  - Investigational Site - Getafe, Getafe
  - Investigational Site - Madrid 1, Madrid
  - Investigational Site - Madrid 2, Madrid
  - Investigational Site - Madrid 3, Madrid
  - Investigational Site - Santiago de Compostela, Santiago de Compostela
  - Investigational Site - Valencia, Valencia

REFERENCES:
- See also: Related Info — http://www.cerexa.com